CLINICAL TRIAL: NCT01267487
Title: Phase 4 Study of Fixed-dose and Titration Schemes of Heparin and Protamine in Cardiopulmonary Bypass Cardiac Surgeries : Evaluation of Post-operatory Blood Loss and Transfusion Requirements
Brief Title: Clinical Trial Comparing Heparin and Protamine Fixed and Titrated Doses in Cardiac Surgery With Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SANE-Society of Anesthesiology (Other)
Collaborators: Instituto de Cardiologia do Rio Grande do Sul (Other); Fundação Universitária de Cardiologia (University Foundation of Cardiology) (Unknown)
Responsible Party: Maria Beatriz Couto Chuquer, CET/ SBA - SANE
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: UP 4316/09
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Anticoagulation
Keywords: Heparin; Protamine; Cardiopulmonary Bypass; Titration
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fixed doses plus PO protamine (Active Comparator): Intraoperative fixed dose schemes (as in "fixed doses plus placebo" group) plus continuous infusion of 25mg/hour of protamine during first 6 PO hours
  Interventions: Drug: Heparin fixed doses; Drug: PO continuous infusion of Protamine
- Titrated doses plus PO protamine (Active Comparator): Same as "titrated doses" arm, plus continuous infusion of 25mg/ hour of protamine during first 6 PO hours
  Interventions: Drug: PO continuous infusion of Protamine; Drug: Heparin and protamine titration
- Fixed doses plus placebo (No Intervention): Before CPB, fixed heparin dose of 400 Units per kg of body weight to achieve an Activated Coagulation Time (ACT) > 480 seconds.
  Reversal of heparin after CPB using 1 : 1 ratio (1 mg of protamine for each 100 units (1mg) of heparin), plus 0.8 mg/kg of protamine at the end of the surgery.
  Continuous infusion of placebo (saline 0.9%) during the first 6 PO hours.
  Interventions: Drug: Heparin fixed doses
- Titrated doses plus placebo (Active Comparator): Titrated doses of heparin before and during CPB and reversal with protamine after CPB calculated by the construction of individualized Bull's dose-response curve.
  Continuous infusion of placebo (saline 0.9%) during first 6 PO hours.
  Interventions: Drug: Heparin and protamine titration

INTERVENTIONS:
Drug: Heparin fixed doses — Fixed doses of 400 units/ kg of patient's body weight before CPB to achieve an ACT > 480 sec. Supplemental doses of 50mg of heparin if ACT <480 sec during CPB.
  Reversal doses of protamine in a 1:1 ratio (1mg of protamine for every mg of heparin administered), plus 0.8mg/kg of protamine at the end of the surgery.
  Arms: Fixed doses plus PO protamine; Fixed doses plus placebo
Drug: PO continuous infusion of Protamine — 25mg/hour in IV continuous infusion during first 6 PO hours
  Arms: Fixed doses plus PO protamine; Titrated doses plus PO protamine
Drug: Heparin and protamine titration — Titrated doses of heparin during CPB were manually calculated using Bull´s dose-response curve, which was based in periodic assessment of Activated-Coagulation Times (ACT)- baseline ACT, after 2mg/kg of heparin at cannulation and every 15 to 30 minutes during CPB.
  Reversal doses of protamine were calculated as a 1:1 ratio of the actual estimated heparin concentration (in mg/kg) at the end of CPB, using the Bull´s dose response curve.
  Arms: Titrated doses plus PO protamine; Titrated doses plus placebo

SUMMARY:
There are currently several schemes described for anticoagulation with heparin and its reversal with protamine during cardiac surgery with CPB. The oldest, and most used in our routine environment, is the scheme of fixed doses, in which a bolus dose of heparin at the start of CPB is established in IU/kg of body weight and the dose of protamine at the end of CPB is calculated based on the initial dose of heparin administered.

These schemes do not take into account the variability inter-patients and can result in overdose or sub-doses of one or both drugs.

The titration schedule of doses of heparin and protamine through the principle of dose-response curve of Bull promotes individualization of dosage according to the response of each patient. This scheme has been associated with an effective reversal of the effect of heparin after CPB and with reduction of post-operatory bleeding and transfusion.

The restoration of a state of anticoagulation by heparin after its reversal by protamine is called "rebound effect". It is a phenomenon explained by the recirculation of heparin stored in the reticulum-endothelial system and connective tissue, or by free residual concentration of heparin after clearance of protamine. This effect may be present for more than 6 hours of post-operatory and may contribute to increase post-operatory bleeding.

DETAILED DESCRIPTION:
The objectives were, primarily, to compare intraoperative fixed versus titrated doses of heparin and protamine in cardiac surgeries with CPB regarding blood loss and transfusion requirements during the first 24 post-operative (PO) hours.

Secondarily, the investigators compared continuous infusion of small doses of protamine (25mg/hour) and placebo during the first 6 PO hours to neutralize heparin rebound effect. The investigators measured KTTP and fibrinogen levels during the first 24 PO hours and also the difference in blood loss and transfusion requirements between the groups.

The study included patients from 18 to 75 years-old submitted to Cardiac surgeries with Cardiopulmonary Bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to an Elective Cardiac Surgery with Cardiopulmonary Bypass
* Age 18 to 75 years-old

Exclusion Criteria:

* Hematocrit < 30
* INR > 1,3
* Platelets < 100,000
* Altered KTTP
* Receiving Non-fractioned Heparin or Low-Molecular Weight Heparin
* Renal Insufficiency or Creatinine > 2,0
* Liver Failure or altered ALT/AST
* Von Willebrands'disease, Haemophilia, sepsis
* Use in the past 7 days of antiplatelet-therapy(Ticlopidine or Clopidogrel)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Mediastinal blood drainage (ml) | First 24 PO hours
  The mediastinal blood drainage was measured hourly during the first 6 post-operatory (PO) hours, and every 6 hours from the 7th to 24th PO hours.

SECONDARY OUTCOMES:
Transfusion of blood components | First 24 PO hours
  We measured the incidence(%) of transfusion of Packed Red Blood Cells, Plasma or Platelet during first 24 PO hours

CONTACTS AND LOCATIONS:
Overall Officials: Maria B Chuquer, M. D., Principal Investigator — SANE-Society of Anesthesiology
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Shore-Lesserson L, Reich DL, DePerio M. Heparin and protamine titration do not improve haemostasis in cardiac surgical patients. Can J Anaesth. 1998 Jan;45(1):10-8. doi: 10.1007/BF03011985. PMID 9466020
- [Background] Teoh KH, Young E, Blackall MH, Roberts RS, Hirsh J. Can extra protamine eliminate heparin rebound following cardiopulmonary bypass surgery? J Thorac Cardiovasc Surg. 2004 Aug;128(2):211-9. doi: 10.1016/j.jtcvs.2003.12.023. PMID 15282457
- [Background] Pappalardo F, Franco A, Crescenzi G, De Simone F, Torracca L, Zangrillo A. Anticoagulation management in patients undergoing open heart surgery by activated clotting time and whole blood heparin concentration. Perfusion. 2006 Dec;21(5):285-90. doi: 10.1177/0267659106074770. PMID 17201083
- [Background] Griffin MJ, Rinder HM, Smith BR, Tracey JB, Kriz NS, Li CK, Rinder CS. The effects of heparin, protamine, and heparin/protamine reversal on platelet function under conditions of arterial shear stress. Anesth Analg. 2001 Jul;93(1):20-7. doi: 10.1097/00000539-200107000-00005. PMID 11429331
- [Background] Bull BS, Huse WM, Brauer FS, Korpman RA. Heparin therapy during extracorporeal circulation. II. The use of a dose-response curve to individualize heparin and protamine dosage. J Thorac Cardiovasc Surg. 1975 May;69(5):685-9. PMID 1127967
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454
- [Background] Jobes DR, Aitken GL, Shaffer GW. Increased accuracy and precision of heparin and protamine dosing reduces blood loss and transfusion in patients undergoing primary cardiac operations. J Thorac Cardiovasc Surg. 1995 Jul;110(1):36-45. doi: 10.1016/S0022-5223(05)80007-8. PMID 7609566
- [Background] Levy JH, Tanaka KA. Anticoagulation and reversal paradigms: is too much of a good thing bad? Anesth Analg. 2009 Mar;108(3):692-4. doi: 10.1213/ane.0b013e31819614dd. No abstract available. PMID 19224768
- [Background] Despotis GJ, Joist JH, Hogue CW Jr, Alsoufiev A, Kater K, Goodnough LT, Santoro SA, Spitznagel E, Rosenblum M, Lappas DG. The impact of heparin concentration and activated clotting time monitoring on blood conservation. A prospective, randomized evaluation in patients undergoing cardiac operation. J Thorac Cardiovasc Surg. 1995 Jul;110(1):46-54. doi: 10.1016/S0022-5223(05)80008-X. PMID 7609568
- [Background] Lobato RL, Despotis GJ, Levy JH, Shore-Lesserson LJ, Carlson MO, Bennett-Guerrero E. Anticoagulation management during cardiopulmonary bypass: a survey of 54 North American institutions. J Thorac Cardiovasc Surg. 2010 Jun;139(6):1665-6. doi: 10.1016/j.jtcvs.2010.02.038. Epub 2010 Mar 19. No abstract available. PMID 20303507